CLINICAL TRIAL: NCT07035158
Title: A Case Control Study in a Population With Clinical Suspicion of Liver Cirrhosis to Develop a Risk Model for the Presence of Cirrhosis Using Breath Biomarkers/EVOC Probes
Brief Title: DELIVER Study in a Population With Clinical Suspicion of Liver Cirrhosis
Acronym: DELIVER
Status: Recruiting | Type: Observational
Sponsor: Owlstone Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: DEL001
Record Dates: First submitted 2024-05-21; First posted 2025-06-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EVOC probe: After confirming full eligibility, the EVOC probe will be administered orally to both cases (individuals with cirrhosis) and controls (individuals with a clinical suspicion of cirrhosis)
  Interventions: Diagnostic Test: Libra Oral Solution

INTERVENTIONS:
Diagnostic Test: Libra Oral Solution — EVOC Probe

SUMMARY:
Owlstone Medical has demonstrated that the use of an Exogenous Volatile Organic Compound (EVOC) that targets specific metabolic processes linked to cirrhosis pathophysiology enables identification of subjects with cirrhosis with high accuracy compared to healthy controls. This approach relies on the oral administration of food additives that are metabolized in the liver resulting in volatile end-products exhaled in breath. The presence of liver cirrhosis alters the metabolism of these EVOC-probes altering the breath concentrations of the end-products. These alterations can be used to identify subjects who have a risk of having liver cirrhosis.

The study is designed as a case control study comparing subjects with cirrhosis against controls originating from a group of subjects with clinical suspicion of cirrhosis. Adequate balancing of subjects across definitive, probable, possible, and absent cirrhosis groups will be assured through a recruitment enrichment strategy. The primary output of the study will be an algorithm to calculate a risk score for the presence of cirrhosis. As a secondary objective sensitivity analysis will be performed to assess the impact of subject characteristics and cirrhosis etiology on test performance to assure robustness of the test in a deployment setting. The results of this study will inform test optimization for a prospective clinical validation trial, with the goal of developing a test that is widely applicable and available in primary care centers

DETAILED DESCRIPTION:
Liver disease and cirrhosis specifically is an area of growing public health concern with serious liver disease frequently presenting at advanced stages. Up to 75% of patients with cirrhosis receive their first diagnosis after they arrive at the accident and emergency department with a failing (decompensating) liver. This late diagnosis can lead to poor prognosis as treatments available are less effective at preserving the liver.

At present early detection is difficult as early disease often has few or no symptoms, and current diagnostic methods are either invasive or have limited accuracy. There is therefore an unmet need for easy to use, non-invasive tests that can help to diagnose cirrhosis earlier, when treatments are still effective at preserving liver function and increasing life expectancy. A breath test may fulfil such requirements.

The DELIVER study aims to develop a breath test that can identify cirrhosis at an earlier stage.

Recent research has shown that cells inside the body produce substances that end up in the lungs and are breathed out, or 'exhaled' in breath. These studies have shown that those substances may be different if someone is suffering from a particular disease, including liver cirrhosis.

Research has also shown that when we ingest a certain product (referred to as a 'probe') it may be processed differently in the body if you are healthy, compared to if you have a particular disease. This is very similar to different bodies digesting foods in different ways. This difference in processing leads to different types of chemicals being released by the body which would show up on breath as a sign of the presence or absence of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to provide written informed consent.
3. Clinical suspicion of cirrhosis evaluated in the last six months preceding the recruitment into the study.

The presence of clinical suspicion is at the discretion of the (referring) clinician. For reference this will typically be based on (a combination of) the following:

* Risk factors: viral hepatitis, metabolic dysfunction associated steatotic liver disease (MASLD), alcoholic liver disease, primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis, haemochromatosis or combinations of these diseases
* Symptoms: e.g. fatigue, weakness, abdominal pain, nausea, vomiting, loss of appetite, oedema, jaundice, spider angioma, palmar erythema, clubbing, gastrointestinal bleeding or altered blood parameters in a liver function test.

Exclusion Criteria:

1. Interventional treatment for (underlying cause of) cirrhosis aimed at disease modification during the past six months. Any treatment solely focused on symptom/complications management are permissible.
2. Received an investigational medicinal product in the context of a Clinical Trial (CTIMP) during the 28 days prior to administration of the (first) probe.
3. Women who are pregnant or breastfeeding, for women of childbearing potential a urine pregnancy test can be administered
4. Known allergy/intolerance to any of the constituents of the EVOC-probe cocktail, specifically limonene, 2-butanol, 2-pentanone, polysorbate 80 (aka Tween-80), and sucralose.
5. Subjects on peritoneal- or hemo-dialysis
6. Primary referral for evaluation of the presence of liver cancer (e.g. abnormal findings on imaging).
7. The presence of histopathologically diagnosed liver cancer.
8. (Anticipated) inability to complete the breath sampling procedure due to e.g., inability to maintain adequate ventilation unaided / Inability to comply with the study procedures in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects that have a clinical suspicion or diagnosis of cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Developing a model to determine the risk of the presence of liver cirrhosis. | 10 months
  The primary objective is to develop a model for determining the risk of the presence of liver cirrhosis based on breath biomarkers and anthropometric factors in a population comprising individuals at risk of liver cirrhosis warranting expert diagnostic evaluation. This will be a cross validated risk model reporting likelihood of the presence of cirrhosis. Model performance will be evaluated using AUC, specificity, sensitivity, NPV, PPV negative and positive likelihood ratios.

SECONDARY OUTCOMES:
Sensitivity Analysis | 10 months
  Perform sensitivity analysis of the risk model for different cirrhosis etiology, and clinical characteristics
Definition of the optimal breath collection method and timepoints | 10 months
  Define the test: Select optimal breath collection method and timepoint(s). An optimal test protocol is identified balancing diagnostic accuracy and acceptability of the breath test protocol to healthcare providers and patients
Correlation of Risk Score | 10 months
  Correlation of risk score with existing tests and methods used to evaluate liver fibrosis stage, if available. Using established diagnostic approaches and risk scores including but not limited to Child Pugh score, MELD, UKELD, FIB4, APRI, liver biopsy parameters, liver stiffness and liver fat, signs of portal hypertension, fibrosis scoring, GGT, ALP, and their individual parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Shankar, Principal Investigator — Norfolk & Norwich University Hospital
Locations (4):
- Arizona Liver Health, Chandler, Arizona, United States
- Hospital Padre Hurtrado, Santiago, Chile
- United Kingdom (2):
  - Norfolk and Norwich Hospital, Norwich
  - Peterborough City Hospital, Peterborough

IPD SHARING:
Plan to Share IPD: No